CLINICAL TRIAL: NCT02335073
Title: Effect of 4 Liver Fibrosis Tests (PIIINP, CIV, LN, and HA) on the Prognosis of Liver Cirrhosis: A Single-center, Prospective, Observational Study
Brief Title: Effect of 4 Liver Fibrosis Tests (PIIINP, CIV, LN, and HA) on the Prognosis of Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Dr., General Hospital of Shenyang Military Region
Other Study IDs: LFT4-LC
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Liver Cirrhosis
Keywords: Prognosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Venous Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Venous blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Venous blood

SUMMARY:
Liver biopsy is the reference method for the measurement of liver fibrosis. But it has many limitations, such as sampling error and individual variation in interpreting the results. Currently, serum liver fibrosis markers have been employed as non-invasive diagnosis of liver fibrosis and evaluation of the severity of liver fibrosis. They include laminin (LN), hyaluronic acid (HA), collagen type IV (CIV), and N-terminal propeptide of collagen III (PIIINP). However, few study was conducted to explore the role of these liver fibrosis markers in evaluating the prognosis of liver cirrhosis. Our hypothesis is that LN, HA, CIV, and PIIINP in combination or alone can predict the prognosis of liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were admitted to our department.
2. Patients were diagnosed with liver cirrhosis.
3. Patients signed the informed consent and agreed to test serum liver fibrosis markers (PIIINP, CIV, LN, and HA).

Exclusion Criteria:

1. Non-cirrhotic patients.
2. Malignancy.
3. Severe cardiopulmonary diseases.
4. Severe infectious diseases.
5. Other diseases with a shortened lifespan.
6. Pregnant and breastfeeding.
7. Poor adherence.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population should be patients with a diagnosis of liver cirrhosis who were admitted to the Department of Gastroenterology of the General Hospital of Shenyang Military Area.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Death | 6-12 months

SECONDARY OUTCOMES:
Hepatic decompensation events | 6-12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, General Hospital of Shenyang Military Area, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No